CLINICAL TRIAL: NCT00525317
Title: Does Oral Magnesium Substitution Relieve Magnesium Induced Leg Cramps ?
Brief Title: Does Oral Magnesium Substitution Relieve Pregnancy Induced Leg Cramps ?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Takeda Nycomed (Unknown); Sykehuset Asker og Baerum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Oral magnesium in pregnance
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Cramps
Keywords: Pregnancy; Magnesium; Leg Pain
MeSH Terms: conditions — Muscle Cramp

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium tablet suplementation (1) (Active Comparator): Nycoplus Magnesium" (120 mg x 3 daily for 2 weeks)
  Interventions: Drug: "Nycoplus Magnesium" (120 mg x 3 daily for 2 weeks)
- Placebo tablet suplementation (2) (Placebo Comparator): Placebo (3 times daily for 2 weeks)
  Interventions: Drug: "Nycoplus Magnesium" (120 mg x 3 daily for 2 weeks)

INTERVENTIONS:
Drug: "Nycoplus Magnesium" (120 mg x 3 daily for 2 weeks) — 120 mg x 3 or placebo
  Other Names: Nycoplus Magnesium tablets(R); Placebo tablets

SUMMARY:
This is a trial of treatment with tablets containing magnesium for leg cramps in pregnancy.

DETAILED DESCRIPTION:
Healthy pregnant women between 18 and 36 weeks of pregnancy suffering from leg cramps at least twice a week were treated with magnesium tablets or placebo for two weeks, 120 mg x 3 daily.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with recurrent leg cramps (at least twice a week).
* No disease according to helath certificate. Written participation consent must be signed.
* Linguistic ability demanded: Norwegian as the first language. Gestation length more than 17 weeks, less than 36 weeks.

Exclusion Criteria:

* Twin pregnancy.
* Oedema.
* Pre-eclampsia.
* Magnesium supplementation beyond the trial treatment.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2002-01; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity and frequency | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bohmer, MD, Principal Investigator — Aker Universituy Hospital